CLINICAL TRIAL: NCT02505230
Title: Meal Presentation and Liking
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: UTK IRB-15-02349-XP
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Volume; Energy Density; Meal Presentation
MeSH Terms: interventions — Eating

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Meal Order 1 (Experimental): [P,P+S,HVP,LVP]
  For the PASTA (P) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) and no vegetables.
  For the PASTA+SIDE (P+S) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) with a side of mixed zucchini and squash (cut in 1/2 inch half-moon slices).
  For the HIGH-VOLUME PASTA (HVP) condition, participants view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) mixed with zucchini and squash (cut in 1/2 inch half-moon slices).
  For the LOW-VOLUME PASTA (LVP) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) mixed with grated zucchini and squash (chopped in food processor).
  Interventions: Behavioral: Eating
- Meal Order 2 (Experimental): [P+S,HVP,LVP,P]
  For the PASTA+SIDE (P+S) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) with a side of mixed zucchini and squash (cut in 1/2 inch half-moon slices).
  For the HIGH-VOLUME PASTA (HVP) condition, participants view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) mixed with zucchini and squash (cut in 1/2 inch half-moon slices).
  For the LOW-VOLUME PASTA (LVP) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) mixed with grated zucchini and squash (chopped in food processor).
  For the PASTA (P) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) and no vegetables.
  Interventions: Behavioral: Eating
- Meal Order 3 (Experimental): [HVP,LVP,P,P+S]
  For the HIGH-VOLUME PASTA (HVP) condition, participants view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) mixed with zucchini and squash (cut in 1/2 inch half-moon slices).
  For the LOW-VOLUME PASTA (LVP) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) mixed with grated zucchini and squash (chopped in food processor).
  For the PASTA (P) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) and no vegetables.
  For the PASTA+SIDE (P+S) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) with a side of mixed zucchini and squash (cut in 1/2 inch half-moon slices).
  Interventions: Behavioral: Eating
- Meal Order 4 (Experimental): [LVP,P,P+S,HVP]
  For the LOW-VOLUME PASTA (LVP) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) mixed with grated zucchini and squash (chopped in food processor).
  For the PASTA (P) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) and no vegetables.
  For the PASTA+SIDE (P+S) condition, participants will view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) with a side of mixed zucchini and squash (cut in 1/2 inch half-moon slices).
  For the HIGH-VOLUME PASTA (HVP) condition, participants view, consume, and evaluate a main pasta entree (Fettuccini Alfredo) mixed with zucchini and squash (cut in 1/2 inch half-moon slices).
  Interventions: Behavioral: Eating

INTERVENTIONS:
Behavioral: Eating — Participants will have 20 minutes to eat as much or as little of a meal (consisting of pasta alone or pasta with zucchini and squash presented in 3 different ways)

SUMMARY:
This study will investigate the energy consumed from an entree with high- or low-volume vegetables incorporated into the entree or served along side of the entree, in normal weight adults.

DETAILED DESCRIPTION:
Participants will complete four experimental sessions, where a main entree with high- or-low volume vegetables (either added as a side item or mixed with the main entree) will be served for lunch, to determine the impact that presentation and liking may have on the consumption of energy dense foods.

Once screened participants arrive for their first experimental session, they will record the foods and beverages they consumed in the past 24 hours, as well as write down the minutes of physical activity they participated in, within that same 24 hour period. The participants will rate their hunger, fullness, and liking of foods using a 100 mm VAS. After completing these forms, participants will be presented the appropriate meal, for their condition. Following the presentation of the meal, the participant will rate their liking of the meal appearance and then be instructed to eat as much or as little as they want of the meal provided in 20 minutes. At the completion of the allotted time, the meal will be removed, and the participant will evaluate their level of hunger, fullness, and liking of the foods consumed. The session will conclude with the collection of the hunger, fullness, and liking forms.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 to 24.9 kg/m^2
* Unrestrained eater (<12 on Three Factor Eating Questionnaire [TFEQ])
* Report liking Fettucini Alfredo, zucchini, and squash (rate all items >50mm on a visual analogue scale [VAS])
* Report regularly eating before 10 am
* Can compete all sessions within 8 weeks of the screening session

Exclusion Criteria:

* Report binge eating
* Report a medical condition that influences eating
* Report allergies to foods used in the investigation
* Currently smoke
* Report dietary restrictions
* Report taking a medication that affects appetite
* Report being pregnant or breast-feeding
* Report being an athlete in training

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Grams of main pasta entree consumed | 20 minutes
Grams of zucchini and squash consumed | 20 minutes
Level of hunger | baseline
Level of fullness | baseline
Level of liking | baseline
Energy intake | 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee, United States

REFERENCES:
- [Background] Rolls BJ, Drewnowski A, Ledikwe JH. Changing the energy density of the diet as a strategy for weight management. J Am Diet Assoc. 2005 May;105(5 Suppl 1):S98-103. doi: 10.1016/j.jada.2005.02.033. PMID 15867904
- [Background] Rolls BJ. The relationship between dietary energy density and energy intake. Physiol Behav. 2009 Jul 14;97(5):609-15. doi: 10.1016/j.physbeh.2009.03.011. Epub 2009 Mar 20. PMID 19303887
- [Background] Rolls BJ, Meengs JS, Roe LS. Variations in cereal volume affect the amount selected and eaten for breakfast. J Acad Nutr Diet. 2014 Sep;114(9):1411-6. doi: 10.1016/j.jand.2014.01.014. Epub 2014 Mar 19. PMID 24656953
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Background] Lohman TR, Roche AF, Martorell R. Anthropometric Standardization Reference Manual. Champaign,Illinois: Human Kinetics Books; 1988.